CLINICAL TRIAL: NCT02934360
Title: Evaluation of the TR(ACE) Assay for the Ability to Aid in Monitoring Disease Progress, Response to Therapy or for Recurrent or Residual Disease for Patients With Previously Diagnosed Cancers (Stage III and IV Lung and Stage IV Breast)
Brief Title: TR(ACE) Assay Clinical Specimen Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biological Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: BioDyn-15-003
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Breast Neoplasms
Keywords: Lung Cancer; Breast Cancer; cell free DNA; biomarker
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma specimens will be collected prospective and tested retrospectively
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-small cell Lung Cancer: Previously diagnosed stage III or higher non-small cell lung cancer subjects will provide serial plasma specimens and clinical assessment information over time
  Interventions: Device: TR(ACE) Assay Testing
- Breast Cancer: Previously diagnosed stage IV breast cancer subjects will provide serial plasma specimens and clinical assessment information over time.
  Interventions: Device: TR(ACE) Assay Testing

INTERVENTIONS:
Device: TR(ACE) Assay Testing — Serial plasma testing with TR(ACE) Assay

SUMMARY:
The TR(ACE) Assay is a quantitative in vitro diagnostic test run on the TR(ACE) Instrument intended for the measurement of high molecular weight human DNA from plasma as an aid to monitoring disease progression or response to therapy or recurrent or residual disease.

DETAILED DESCRIPTION:
This study is to establish the clinical performance of the TR(ACE) Assay. Deltas of serial TR(ACE) Assay measurements will be compared to the standard of care physician clinical assessment and RECIST 1.1 criteria evaluation relative to the previous visit. Significant changes in serial TR(ACE) Assay measurements are hypothesized to correlate with disease progression or response.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung: Male or Female Adult patient >= 21 years old
* Breast only: Female Adult patient >= 21 years old
* Previously diagnosed with one of the following cancers:

Breast or Non-small Cell Lung

* Cancer has progressed to at least Stage III or higher for lung cancer or,
* Cancer has progressed to stage IV (metastatic) breast cancer
* Participating in standard of care cancer therapy requiring frequent treatments, typically intravenous chemotherapy visits (or as determined by the standard of care for the particular cancer assessed), of a minimum of three (3) treatment visits planned in 9 months from date of enrollment where a clinical assessment will be conducted

Exclusion Criteria:

* Physician assessment that obtaining two extra whole blood specimens with minimum volume of 5 mL per treatment visit is contraindicated
* Stage I and II Non-small Cell Lung Cancer
* Stage I through III breast cancer
* Pregnant or planning to become pregnant during the course of the study
* Unable to obtain informed consent from subject or their legal representative
* Life expectancy is less than 9 months
* Presence of one or more of the following other chronic diseases
* Another type of cancer except for non-melanomatous skin tumors
* Autoimmune disease requiring DMARDS or Biologics
* Infectious disease requiring prolonged intravenous antibiotics or hospitalization
* Renal disease specifically those in End Stage Renal Failure
* Recent (< 3 weeks) major trauma or major surgical procedure(s) or radiation therapy prior to enrollment in the study
* Recent (< 2 months) major occlusive arterial event such as MI or CVA prior to enrollment in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously diagnosed non-small cell lung cancer subjects undergoing standard of care treatment Previously diagnosed breast cancer subjects undergoing standard of care treatment
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Assessment change | Standard of care (approximately every 6 weeks to 3 months) for 6- 9 months
  Standard of care physician's clinical assessment of disease progression or response compared to previous visit

SECONDARY OUTCOMES:
RECIST 1.1 criteria | Standard of care (approximately every 6 weeks to 3 months) for 6- 9 months
  RECIST 1.1 criteria of subjects from current to previous visit

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kovelman, Study Director — Biological Dynamics
Locations (16):
- United States (16):
  - California Cancer Associates for Reseach and Excellence, Inc. (cCare), Encinitas, California
  - North County Oncology Medical Inc. (North County), Oceanside, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Mid-Florida, Orange City, Florida
  - Bond Clinic, Winter Haven, Florida
  - Indiana University Health Bloomington, Bloomington, Indiana
  - Ashland Bellefonte Cancer Center, Ashland, Kentucky
  - Michmer (Lake Huron Medical Center), Port Huron, Michigan
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - North Shore Hematology Oncology, East Setauket, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - AnMed, Greenville, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Tyler Hematology Oncology, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Following direct de novo submission, data will be summarized in decision summary and package insert